CLINICAL TRIAL: NCT01376401
Title: Bendamustine, Bortezomib (Velcade ®) and Prednisone (BVP) in Patients Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Mundipharma Pharmaceuticals B.V. (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BenVelPres
Record Dates: First submitted 2011-06-15; First posted 2011-06-20 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Bortezomib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bendamustine
Drug: Velcade
Drug: Prednisone

SUMMARY:
This protocol corresponds to an open-label national phase II, multicenter, to assess efficacy (in terms of response rate and CR) and toxicity of bendamustine, bortezomib and prednisone (BVP) in 60 patients newly diagnosed MM. Patients in the absence of disease progression or unacceptable toxicity receive up to 9 cycles of BVP. The patients eligible for autologous transplant receive four cycles of BVP, hematopoietic stem cell collection and administration of two cycles BVP over followed by autologous transplant.

In addition to the overall response rates, will also be analyzed time to progression (TTP), progression-free survival (PFS) and overall survival.

Finally, the results will be compared with BVP with those obtained in 120 patients included in our protocol VMP GEM10MAS65.

Patients will be evaluated at scheduled visits up to 3 periods of study:

pretreatment, treatment and monitoring.

DETAILED DESCRIPTION:
Patients included in the study will receive a 6 week cycle consisting of Bendamustine administered IV at doses of 90 mg/m2 on days 1 and 4 of the first cycle and days 1 and 8 in subsequent cycles in combination with Bortezomib as a bolus dose of 1.3 mg/m2 on days 1, 4, 8, 11, 22, 25, 29 and 32, and oral prednisone at doses of 60 mg/m2, during the first four days of each cycle.

Then, patients will receive eight additional cycles of 5-week . The same pattern consisting of bendamustine and prednisone but bortezomib is administered as an intravenous bolus dose of 1.3 mg/m2 on days 1, 8, 15 and 22.

ELIGIBILITY:
Inclusion Criteria:

* Patient age greater than or equal to 18 at the time of signing Informed consent
* Patient who has voluntarily signed informed consent before conduct of the trial any evidence that is not part of care normal patients, with the knowledge of the patient that can leave the trial at any time he want
* Patient able, in the opinion of the physician to comply with the visitation schedule and other requirements of the protocol
* Patient newly diagnosed symptomatic multiple myeloma based on standard criteria and has not received any previous treatment of chemotherapy for MM.
* Patients with newly diagnosed multiple myeloma, secretory, or oligosecretor or not secretor if it has soft tissue plasmacytomas.
* Patients with non-secretory MM oligosecretor or without white tissue plasmacytomas be excluded to keep a group of patients with characteristics similar to the previous study with which we compare the results.
* Patients with measurable disease, defined by the following criteria:

For MM secreting measurable disease is defined as any value quantifiable serum monoclonal protein (≥ 1g/dl) and where applicable, a light chain excretion in urine ≥ 200 mg/24 hours. For Multiple Myeloma oligosecretor or secreting measurable disease defined by the presence of soft tissue plasmacytomas (not bone) determined by clinical examination or radiographic methods (eg MRI, CT-Scan)

* ECOG PS ≤ 2
* Expectations of life than 3 months.
* The patient has the following laboratory values within 28 days before the baseline visit:

Platelet count ≥ 100 x 109 / L, hemoglobin ≥ 8.0g/dL and absolute neutrophil count (ANC) ≥ 1.5 x 109 / L; allowed counts under if they are clearly due to a bone marrow infiltration by MM.

Corrected serum calcium <14mg/dL. Aspartate transaminase (AST) ≤ 2.5 x upper limit of normal(LSN) Alanine aminotransferase (ALT) ≤ 2.5 x ULN Total bilirubin within normal limits Serum creatinine <2 mg / dL

- Patients of childbearing potential must use effective contraception during duration of the study and up to 6 months after completion of treatment

Exclusion Criteria:

* Patient has previously received treatment for multiple myeloma with Pulse steroids except for some emergency that requires it before start of induction therapy, administration of bisphosphonates or radiation therapy, or analgesic due to the presence of plasmacytomas, which require it for some urgency.
* Patients with non-measurable disease.
* Patient with peripheral neuropathy grade ³ 2 within 14 days prior to its inclusion in the trial
* Patients with hypersensitivity to bortezomib, boric acid, or bendamustine mannitol
* Patient to be known carrier of the virus HIV (human immunodeficiency) surface antigen of hepatitis B virus or who has active infection virus hepatitis C.
* Patient who has had a myocardial infarction within 6 months prior to inclusion in the clinical trial or has a functional class III or IV according to the New York Heart Association (NYHA) heart failure, uncontrolled angina, uncontrolled ventricular arrhythmias or acute ischemia detected electrocardiographically or conduction system disorders.
* Patient who has received any investigational agent within 30 days prior their inclusion or is currently in another clinical trial or receiving any investigational agent
* Patient undergoing major surgery within 30 days before inclusion in the study
* Patient pregnant or breastfeeding
* Patients with acute diffuse infiltrative pulmonary disease and / or disease pericardium
* History of other malignancies after different myeloma (except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) to unless the patient is free of the disease beyond 5 years
* Hypertension arterial or poorly controlled diabetes mellitus or any other disease severe organ involving an unreasonable risk to the patient
* Any psychiatric disorder that interferes with comprehension of consent informed or prevent the normal discharge that requires participation in this trial
* Patients with major psychiatric history.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of response rate and complete response rate (CR and near CR) | 1 year

SECONDARY OUTCOMES:
Safety in terms of toxicity | 1 year
Time to progresion | 3 years
Progresion free survival | 2 years
Global survival | 3 years

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínic, Barcelona
  - Institut català d'Oncología, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson Internacional, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Morales Messeguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Mateos MV, Oriol A, Rosinol L, de Arriba F, Puig N, Martin J, Martinez-Lopez J, Echeveste MA, Sarra J, Ocio E, Ramirez G, Martinez R, Palomera L, Payer A, Iglesias R, de la Rubia J, Alegre A, Chinea AI, Blade J, Lahuerta JJ, San Miguel JF. Bendamustine, bortezomib and prednisone for the treatment of patients with newly diagnosed multiple myeloma: results of a prospective phase 2 Spanish/PETHEMA trial. Haematologica. 2015 Aug;100(8):1096-102. doi: 10.3324/haematol.2015.124818. Epub 2015 Apr 24. PMID 25911554
- See also: Spanish Association of Hematology — http://aehh.org